CLINICAL TRIAL: NCT00378365
Title: A Randomized Trial Assessing the Role of Arsenic Trioxide and/or ATRA During Consolidation Course in Newly Diagnosed Acute Promyelocytic Leukemia (APL)
Brief Title: Acute Promyelocytic Leukemia 2006 (APL)
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: P050604
Record Dates: First submitted 2006-09-18; First posted 2006-09-20 (Estimated); Last update posted 2014-04-16 (Estimated); Status verified 2007-03

CONDITIONS: Leukemia, Promyelocytic, Acute
Keywords: Acute promyelocytic leukaemia; ATRA; Idarubicin; Arsenic trioxide; Patient with a newly acute promyelocytic leukaemia (APL); Unmapped MeSH term
MeSH Terms: conditions — Leukemia, Promyelocytic, Acute | interventions — Arsenic Trioxide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- 1 (Experimental): Arsenic trioxide
  Interventions: Procedure: Arsenic trioxide; Procedure: ATRA

INTERVENTIONS:
Procedure: Arsenic trioxide — Arsenic trioxide
Procedure: ATRA — ATRA

SUMMARY:
To assess the role of Arsenic trioxide and/or ATRA during consolidation course in APL. It is hoped that the investigational arms will further increase the event-free survival at 2 years, with reduced toxicity and without increasing the relapse rate by comparison with a classical anthracycline-AraC consolidation regimen.

DETAILED DESCRIPTION:
Definition: Extended description of the protocol, including information not already contained in other fields, such as comparison(s) studied.

APL is a specific type of acute myeloid leukemia (AML) characterized by its morphology (M3 or M3v in the FAB classification), t(15;17) translocation leading to PML-RARa fusion gene, and by a specific coagulopathy combining D.I.C., fibrinolysis and non specific proteolysis. ATRA can differentiate APL blasts in VITRO and in vivo. The combination of ATRA and anthracycline based chemotherapy yields CR rates greater than 90% in newly diagnosed APL. With early introduction of anthracycline AraC chemotherapy during induction treatment, and maintenance combining continuous 6MP and MTX to intermittent ATRA, the relapse risk in APL therefore now appears to be in the range of 10 to 15%.

Nevertheless, 5 to 10% of the patients do not achieve CR and 10% to 15% still relapse. Another subset of patients (5 to 7% in APL 93 trial including 17% of patients aged greater than 65 years) die in CR, from complications of the consolidation treatment phase, mainly from infection during chemotherapy induced aplasia. Failure to achieve CR with current treatment approaches is almost exclusively due to early death during induction treatment. Causes of death are predominantly bleeding, ATRA syndrome and less often infection. Early deaths predominate in elderly patients and patients with high WBC counts. Reducing the amount of chemotherapy administered to newly diagnosed APL patients diminishes this toxicity. The Spanish PETHEMA group reported results of two successive phase II trials in newly diagnosed APL with ATRA and chemotherapy with intercalating agents (idarubicin and mitoxantrone) without AraC followed by maintenance combining ATRA and low dose chemotherapy (LPA96 and LPA99 trials). Results appeared similar to those of the best arm of APL 93 trial, but with less toxicity and only 2 to 3 % death in CR were seen, including in elderly patients.

Arsenic trioxide (As2O3 or ATO) is an effective agent in relapsing or refractory APL, which induced 85% hematological and 79% molecular CR rates in a pivotal US study. The interest of ATO in the front-line therapy of newly-diagnosed APL has been strongly suggested in three studies which showed high complete remission rate, low incidence of relapse and limited toxicity.

In this study, patients will be stratified based on age (≤ 70 years and > 70 years) and WBC count at diagnosis (WBC<10.000/mm3 and >10.000 /mm3).

-Patients aged 70 years or less with WBC<10.000/mm3.

In this population (about 70 % of APL) the best treatment group of APL2000 trial (ATRA with early introduction of anthracycline-AraC chemotherapy but where Idarubicin will be substituted for Daunorubicin, followed by 2 anthracycline-AraC consolidation courses and maintenance combining continuous chemotherapy and intermittent ATRA) will be compared to the same regimen, but without AraC during consolidation courses which will be replaced by:

* either ATO
* or ATRA It is hoped that the investigational arms will further increase the event-free survival at 2 years, with reduced toxicity and without increasing the relapse rate by comparison with a classical anthracycline-AraC consolidation regimen.

  * Patients aged 70 years or less with WBC>10.000/mm3 Patients ages 70 years or less with initial WBC counts > 10000/mm3 (ie very high counts for APL), which represent about 20% of APL, remain at relatively high risk of relapse even with the current reference treatment. The main objective of the study will be to test the addition of ATO during consolidation courses to our current standard ATRA and chemotherapy regimen. Patients will receive the best treatment group of APL 2000 trial (but where Idarubicin will be substituted for Daunorubicin) with or without ATO during the 2 consolidation cycles.
  * Patients older than 70 years with WBC<10.000 /mm3. Elderly patients with initial WBC ≤ 10000/m3 (about 8% of APL) and no contra indication to this treatment will receive a regimen with reduced cumulative dose of chemotherapy but addition of ATO during consolidation courses and during the first year of maintenance treatment. The main purpose of this non randomized part of the trial is to reduce the early death mortality and death in CR observed in elderly patients, without increasing the relapse rate.
  * Patients older than 70 years with WBC>10.000 /mm3. Elderly patients with initial WBC > 10000/m3 (about 2 to 3% of APL) and no contra indication to intensive regimen will receive the same regimen as those with low WBC but with moderate doses of Aracytine during the induction and during the first consolidation course. The main purpose of this non randomized part of the trial is to reduce the early death mortality and death in CR observed in elderly patients, without increasing the relapse rate.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of APL based on morphological grounds, which will have to be confirmed by the presence of t(15;17) and/or PML-RARA rearrangement with characterization of the bcr subtype (PML-RAR characterization).
* Untreated patients.
* No contraindication to intensive chemotherapy (especially well documented cardiac contraindication to idarubicin).
* In female patients: absence of pregnancy and adequate contraceptive methods (due to teratogenetic effects of ATRA in early pregnancy).
* Absence of Hypersensitivity to Arsenic derivatives.
* No QT interval prolongation or complete atria-ventricular block.
* Written informed consent.

Exclusion Criteria:

* Patients already treated.
* Patients with contraindication to intensive chemotherapy, especially well documented cardiac contraindication to Idarubicin.
* In female patients: pregnancy or absence of adequate contraceptive Methods
* QT interval prolongation or complete atria-ventricular block.
* Hypersensitivity to Arsenic derivatives.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 800 (Estimated)
Dates: Start 2006-10; Primary Completion 2016-09 (Estimated); Study Completion 2016-09 (Estimated)

PRIMARY OUTCOMES:
For Patients aged 70 years or less with WBC<10.000/mm3, The primary end point will be event free survival at 2 years from CR achievement | during de study
  For Patients aged 70 years or less with WBC<10.000/mm3, The primary end point
For patients older than 70 years with WBC>10.000 /mm3, The primary end point will be EFS at 2 years from diagnosis | during the study
  For patients older than 70 years with WBC>10.000 /mm3, The primary end point will be EFS at 2 years from diagnosis

SECONDARY OUTCOMES:
For Patients aged 70 years or less with WBC<10.000/mm3 : | during the study
  For Patients aged 70 years or less with WBC<10.000/mm3 :
Relapse (molecular or hematological). | during the study
  Relapse (molecular or hematological).
Kinetics of decrease of PML-RARA transcript level during and after consolidation course. | during the study
  Kinetics of decrease of PML-RARA transcript level during and after consolidation course.
Survival at 2 years. | during the study
  Survival at 2 years.
Side effects of the treatment, including treatment-related mortality and morbidity of consolidation treatment. | during th study
  Side effects of the treatment, including treatment-related mortality and morbidity of consolidation treatment.
Days on antibiotics, transfusion requirement and nights spent in Hospital | during the study
  Days on antibiotics, transfusion requirement and nights spent in Hospital
For Patients aged 70 years or less with WBC>10.000/mm3 | during the study
  For Patients aged 70 years or less with WBC>10.000/mm3
event free survival at 2 years from CR achievement | during the study
  event free survival at 2 years from CR achievement
Side effects of the treatment, including treatment-related mortality and morbidity of consolidation treatment. | during the study
  Side effects of the treatment, including treatment-related mortality and morbidity of consolidation treatment.
For Patients older than 70 years with WBC<10.000 /mm3 | during the study
  For Patients older than 70 years with WBC<10.000 /mm3
Kinetics of decrease of PML-RARA transcript level during and after consolidation course. | during the study
  Kinetics of decrease of PML-RARA transcript level during and after
Relapse and survival at 2 years. | during the study
  Relapse and survival at 2 years.
Side effects of the treatment, including mortality and morbidity of consolidation treatment. | during the study
  Side effects of the treatment, including mortality and morbidity of
For patients older than 70 years with WBC>10.000 /mm3 | during the study
  For patients older than 70 years with WBC>10.000 /mm3

CONTACTS AND LOCATIONS:
Overall Officials: Lionel ADES, MD,PhD, Principal Investigator — Assistance Publique Hopitaux de Paris
Locations (1):
- Chu Avicenne, Bobigny, France

REFERENCES:
- [Derived] Ades L, Thomas X, Bresler AG, Raffoux E, Spertini O, Vey N, Marchand T, Recher C, Pigneux A, Girault S, Deconinck E, Gardin C, Tournilhac O, Lambert JF, Chevallier P, de Botton S, Lejeune J, Dombret H, Chevret S, Fenaux P. Arsenic trioxide is required in the treatment of newly diagnosed acute promyelocytic leukemia. Analysis of a randomized trial (APL 2006) by the French Belgian Swiss APL group. Haematologica. 2018 Dec;103(12):2033-2039. doi: 10.3324/haematol.2018.198614. Epub 2018 Jul 19. PMID 30026341